CLINICAL TRIAL: NCT01524172
Title: Yoga Based Psychotherapy Group Feasibility and Efficacy Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Harolyn M.E.Belcher, M.D., Director of Research, Family Center at Kennedy Krieger Institute, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00021817
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Emotional Lability; PTSD
Keywords: child trauma exposure; mental health; yoga; mood regulation; child maltreatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Mental Health Treatment (Active Comparator): Trauma-informed evidence supported mental health treatment
  Interventions: Behavioral: Standard Mental Health Treatment
- Yoga Based Psychotherapy Group (Experimental): Yoga Based Psychotherapy will be used as an adjunct mental health interventions
  Interventions: Behavioral: Yoga Based Psychotherapy Group

INTERVENTIONS:
Behavioral: Yoga Based Psychotherapy Group — YBPG promotes self-regulation (attention span and physical and verbal expression/outbursts); self-soothing (breathing and movement techniques that physiologically calm when the child encounters stress or reminders of trauma); competency (successful social interaction, appropriate expression of needs and feelings, healthy coping with stress or crisis); self-awareness (of thoughts and feelings by first increasing awareness of the body and its sensations through yoga); self-esteem (positive self-regard, increase accomplishments and awareness that all individuals have different abilities); and safety and personal boundaries (establishing personal boundaries and respecting others' personal boundaries, differentiate safe and unsafe behaviors and situations).
  Other Names: YBPG
  Arms: Yoga Based Psychotherapy Group
Behavioral: Standard Mental Health Treatment — Trauma and evidence informed therapy
  Arms: Standard Mental Health Treatment

SUMMARY:
This preliminary study will examine the feasibility of conducting a randomized clinical trial of Yoga Based Psychotherapy (YBPG) and standard care mental health (SCMH) treatment compared to SCMH for children ages 8-12 years who have a history of neglect and maltreatment (trauma). The goal of the study is to inform the method and sample size for a larger randomized trial to study the effect of YMBT with SCMH compared to SCMH in improving child regulation of behavior, emotions, and daily functioning. Children who have experienced trauma, including sexual abuse, physical abuse, emotional abuse, exposure to community or domestic violence, parental substance abuse, mental health disorders, and incarceration are at risk to have dysregulation of mood, emotions and behavior. In addition, children exposed to neglect and trauma may have poor attachment to caregivers and poor peer relations. It is hypothesized the using YBPG as an adjunct to SCMH may improve children's regulation of emotion and behavior.

DETAILED DESCRIPTION:
One hundred fifty children (ages 8-12 years) treated at the Center for Child and Family Traumatic Stress (CCTFS) for at least 3 months and their caregivers (total n=300 individuals) will be eligible to be enrolled in this randomized preliminary study if CCTFS Clinician identifies that the child is continuing to have difficulty with behavior and emotional regulation. Children will be invited to participate in the study. Informed consent will be obtained following explanation of the study. If the child meets both Stage 1 and 2 Screening criteria,

Stage 1 Screening:

Child receives a T-score > 60 on any of the Child Behavior Checklist Parent Rating Scales, and

Stage 2 Screening:

KKFC Psychiatric evaluation (Child Psychiatrist will be masked to study status). Child Psychiatrist evaluation will determine whether medication is appropriate for the child and whether the child/family environment is stable and safe. If the child is deemed appropriate for psychotropic medications, other than stimulants, the child will not be eligible for the study (due to the possible changes in one of the outcome measures, heart rate variability, that will likely result from use of psychotropic medications that can not be stopped 24 hours prior to study evaluation). [Children on stimulant medication will be asked to stop medication one day prior to study evaluation and of the day of evaluation.]

The child will be randomized to Group 1: to continue Standard Care Mental Health (SCMH) treatment or Group 2: Standard Mental Health and Yoga Based Psychotherapy Group.

Children with T-scores lower than 60 will continue in Standard Mental Health Treatment. Recruitment will take place over three years.

A block randomization design (block size 4) will be used to ensure roughly equal distribution of YBPG and SCMH patients over the enrollment time. An opaque bag with four colored marbles (two red, two black) will be utilized for the randomization. The child, in the presence of the parent, will be asked to select a colored marble out of the bag; the marbles will be replaced after enrollment of sets of 4 children. Depending on the color of the marble the child will be assigned to either YBPG or SCMH.

Children randomized to YBPG must be cleared by their pediatric care provider (Appendix 1). Children in YBPG group will participate in YBPG as outlined in Appendix 2; participation duration is expected to be 12 weeks. Parents in the YBPG group will participate in a psychoeducational intervention to learn about YBPG and support the child's practice of YBPG. Following 12 weeks of YBPG children will resume SCMH if necessary.

Children will be assessed following informed consent, at 3 months (following YBPG or 6 months of SCMH), 6 months, and 12 months following randomization.

Assessments:

1. Baseline EKG and respiratory rate (RR) will be measured for 5 minutes. Heart rate variability will be measured using a data collection system that will take EKG and respiratory rate recordings for 5 minutes, and analyzed using the CardioBatch software from the Brain Body Center of the University of Illinois. The Trier Social Stress Test 13 for children will be administered. The Trier consists of the research assistant telling the child the beginning of a story and having the child complete the story in 5 minutes. Then the child is asked to perform math problems for 5 minutes. EKG and respiratory rate (RR) will be re-measured for 10 minutes after the Trier.
2. Child Behavior Checklist (CBCL) 14;15. The CBCL is a written measure designed to assess behavioral and emotional problems in children. There are several forms including a version for children from 1 1/2 to 5 years and a version for children 6-18 years 14;15. There are also Parent, Youth, and Teacher rating forms. The Youth Behavior Rating will be used to obtain a self-report of the child's behavioral and emotional status. Each version yields standard scores (Mean = 50, standard deviation = 10) to assess behavior problems in several specific areas; these scores are also combined into three global scores: an Internalizing score for emotional problems, an Externalizing score for behavior problems, and a Total problem score. The Parent Questionnaire form of the CBCL will be used. The CBCL is expected to take 20 minutes to complete.
3. Trauma Symptom Checklist for Young Children (TSCYC) and Trauma Symptom Checklist for Children (TSCC) 16: The TSCYC is a 90-item parent report of children's symptoms associated with traumatic events (e.g., child abuse, peer assaults, community violence). The TSCYC is normed and standardized as a trauma measure for children ages three to 12 years and includes measurements of validity of parent report and norms for the number of waking hours the parent spends with the child during an average week. The instrument includes nine subscales, Post-traumatic Stress-Intrusion, Post-traumatic Stress-Avoidance, Post-traumatic Stress-Arousal, Post-traumatic Stress-Total, Sexual Concerns, Dissociation, Anxiety, Depression, and Anger/Aggression. The TSCYC is expected to take 15-20 minutes to complete. Alpha values on a multi-site clinical sample of traumatized children ranged from 0.81 for Sexual Concerns to 0.93 for Post-traumatic Stress-Total17. The TSCC is a 54 item child questionnaire that has Anxiety, Depression, Anger, Posttraumatic Stress, Dissociation, and Sexual Concerns. Alpha values range from 0.77 for Sexual Concerns to 0.89 for Anger. The TSCC is expected to take 10-15 minutes to complete.
4. Behavior Emotional Rating Scale (BERS-2) 18: The BERS-2 is a 52-item Likert scale that measures the children emotional and behaviors strengths through parent, child, and observer report. The BERS-2 is designed for children ages 5 years to 18 years and is divided into five subscales, namely, (1) Interpersonal Strengths, (2) Family Involvement, (3) Intrapersonal Strengths, (4) School Functioning, and (5) Affective Strengths. Teacher/Clinician, Parent, and Youth Rating Scales will be used in this grant to assess child behavioral and emotional functioning. Cultural/ethnic normative sample were representative of the United States population. Internal consistency ranges from 0.77 to 0.99. The BERS is expected to take 15 minutes to complete.
5. The University of California Los Angeles-Post Traumatic Stress Disorder (UCLA-PTSD) is used to screen both for exposure to traumatic events and for DSM-IV PTSD symptoms in children and adolescents who report traumatic experiences. The UCLA PTSD is expected to take approximately 15 minutes.
6. The Ontario Child Neglect Index (CNI) is a clinician administered assessment designed to identify types and severity of different forms of child neglect. It is designed for use with families already identified by a child protective service agency. The CNI is a 6-scale index and utilizes a 4- to 5-level rating of severity (e.g., adequate, inconsistent, inadequate, seriously inadequate). The score is interpreted as a severity rating of neglect, rather than a binary (yes/no) neglect score. Scores can range from 0-80. The recommended cutoff score is 50. The CNI is expected to take approximately 5 minutes to complete.
7. Demographic information (e.g, gender, age, race/ethnicity, parental age, education, employment, marital status, etc.) will be collected. In addition, medical information including medications, psychiatric diagnosis, birth history, history of maltreatment and psychosocial history will be obtained by parent interview or electronic record review.

ELIGIBILITY:
Inclusion criteria:

* Children, ages 8-12 years,
* enrolled in treatment at KKFC and their caregivers will be invited to participate if the child continues to exhibit behavior dysregulation (Conners' Parent Rating Scale-Revised (S) of > 60) following 3 months of SCMH at the KKFC.
* Children may have a history of receiving psychotropic medications or be currently taking stimulants at the time of study enrollment.

Exclusion criteria:

* Children who are on psychotropic medications or medications that affect their heart rates, other than stimulants will be excluded from this preliminary study.
* Children with cardiac arrhythmias, endocrine disorders associated with heart rate irregularities or who are not able to cooperate or understand study procedures will be excluded.
* Non-English speaking children will be excluded. Children in foster care placements will be excluded.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
To examine the feasibility of recruiting and conducting the proposed intervention and evaluation procedures on a cohort of children exposed to neglect and trauma and their caregivers using a randomized design. | 8 years
  Acceptance rate

SECONDARY OUTCOMES:
Examine the effects of YBMT on heart rate variability, behavior, post traumatic stress disorder symptoms, and functioning. | 8 years
  Improved behavior

CONTACTS AND LOCATIONS:
Overall Officials: Harolyn ME Belcher, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States